CLINICAL TRIAL: NCT00673309
Title: Assessment of Mechanisms of Improved Wound Healing of Anabolic Agents and Diet in Severely Burned Patients
Brief Title: Assessment of Mechanisms of Improved Wound Healing
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00-454; P50GM060338 (NIH); R01GM056687 (NIH); SHC #8660 (Other Grant/Funding Number: Shriners Hospital for children)
Record Dates: First submitted 2007-12-26; First posted 2008-05-07 (Estimated); Results first posted 2019-12-16 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Burns
Keywords: burns
MeSH Terms: conditions — Burns | interventions — Insulin; Oxandrolone; Nandrolone; Propranolol; Growth Hormone; Insulin-Like Peptides; Itraconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- Growth Hormone (Experimental): Growth Hormone administered daily until 95% wound healing. Stable Isotope Infusion Study with collection of blood and tissue
  Interventions: Procedure: Stable Isotope Infusion study; Drug: Growth Hormone
- Insulin High Dose (Experimental): Insulin IV administered continuously to 95% healing. Stable Isotope Infusion Study with collection of blood and tissue
  Interventions: Procedure: Stable Isotope Infusion study; Drug: Insulin High Dose
- Oxandrolone (Experimental): Oxandrolone administered daily until 95% wound healing Stable Isotope Infusion Study with collection of blood and tissue
  Interventions: Procedure: Stable Isotope Infusion study; Drug: oxandrolone
- Propranolol (Experimental): Propranolol administered daily until 95% wound healing Stable Isotope Infusion Study with collection of blood and tissue
  Interventions: Procedure: Stable Isotope Infusion study; Drug: Propranolol
- IGF-1/IGFBP-3 (Experimental): IGF-1/IGFBP-3 will be administered until 95% wound healing
  Interventions: Procedure: Stable Isotope Infusion study; Drug: IGF-1/IGFBP-3
- Insulin Low Dose (Experimental): Insulin Low Dose will be administered until 95% wound healing.
  Interventions: Procedure: Stable Isotope Infusion study; Drug: Insulin Low Dose
- Itraconazole (Experimental): Itraconazole will be administered until 95% wound healing.
  Interventions: Procedure: Stable Isotope Infusion study; Drug: Itraconazole
- Growth Hormone and Propranolol (Experimental): Growth Hormone and Propranolol will be administered until 95% wound healing.
  Interventions: Procedure: Stable Isotope Infusion study; Drug: Growth Hormone and Propranolol
- Oxandrolone and Propranolol (Experimental): Oxandrolone and Propranolol will be administered until 95% wound healing
  Interventions: Procedure: Stable Isotope Infusion study; Drug: Oxandrolone and Propranolol
- Control/Placebo (Placebo Comparator): Placebo or Control will be administered until 95% wound healing
  Interventions: Procedure: Stable Isotope Infusion study; Drug: Placebo or Control

INTERVENTIONS:
Procedure: Stable Isotope Infusion study — Stable isotope infusion study to be done following each surgery. Tagged isotopes to assess uptake into blood and tissues. Includes collection of blood and tissues (muscle)
Drug: Insulin High Dose — Insulin IV administered continuously throughout hospitalization until wounds are 95% healed.
  Other Names: Regular Insulin
  Arms: Insulin High Dose
Drug: oxandrolone — Oxandrolone given daily throughout hospitalization until 95% wound healing.
  Other Names: nandrolone
  Arms: Oxandrolone
Drug: Propranolol — Propranolol to be given daily throughout hospitalization until 95% wound healing.
  Arms: Propranolol
Drug: Growth Hormone — Recombinant Human Growth hormone to be administered daily until 95% wound healing.
  Other Names: GH; rhGH; recombinant human Growth Hormone
  Arms: Growth Hormone
Drug: Insulin Low Dose — Insulin administered IV until 95% wound healing
  Other Names: Insulin
  Arms: Insulin Low Dose
Drug: IGF-1/IGFBP-3 — Insulin Like Growth Factor-1/Insulin like Growth Factor Binding Protein 3 administered until 95% wound healing
  Other Names: Insulin Like Growth Factor
  Arms: IGF-1/IGFBP-3
Drug: Itraconazole — Itraconazole administered until 95% wound healing
  Arms: Itraconazole
Drug: Growth Hormone and Propranolol — Growth Hormone and Propranolol given until 95% wound healing
  Other Names: GH and Propranolol
  Arms: Growth Hormone and Propranolol
Drug: Oxandrolone and Propranolol — Oxandrolone and Propranolol
  Arms: Oxandrolone and Propranolol
Drug: Placebo or Control — Administration of Placebo or Control until 95% wound healing
  Arms: Control/Placebo

SUMMARY:
The purpose of this study is to find ways to improve wound healing and decrease the negative effects of trauma from burn injury.

DETAILED DESCRIPTION:
This study involves research and the investigators hope to learn the following: how or what effect one or more anabolic ("tissue building") agents have on muscle metabolism, wound healing, and immune function after severe burn. The agents include the following: growth hormone, insulin-like growth factor-1 in combination with its binding proteins, insulin, Beta-adrenergic blockers, Alpha Adrenergic Agonist, anabolic steroids such as testosterone, Oxandrolone and nandrolone, ketoconazole and its derivatives, dehydroepiandrosterone, fenofibrate, diet or the application of skin substitute.

ELIGIBILITY:
Inclusion Criteria:

* Patient is between 0 and 90 years of age
* Patient 18 years and older consents to participate in study protocol. If patient is not able to consent, consent will be obtained from closest family member or legal guardian. Parental permission will be obtained for patients less than 18 years of age. Assent will be obtained from children 7-17 years of age if child is physically/mentally able to do so.
* greater than 30% TBSA burn requiring at least 1 operation with donor sites for skin grafting

Exclusion Criteria:

* Known history of AIDS, AIDS-related complex, Human Immunodeficiency Virus
* History of cancer within 5 years
* Tuberculosis, arthritis, cirrhosis, hyperlipidemia, bone or endocrine diseases, autoimmune diseases
* Chronic glucocorticoid or non-steroidal anti-inflammatory drug therapy

Max Age: 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 644 (Actual)
Dates: Start 2000-07; Primary Completion 2011-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David N. Herndon, MD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

REFERENCES:
- [Derived] Zinter MS, Markovic D, Asaro LA, Nadkarni VM, McQuillen PS, Sinha P, Matthay MA, Jeschke MG, Agus MSD, Sapru A; CAF-PINT Investigators of the PALISI Network. Tight Glycemic Control, Inflammation, and the ICU: Evidence for Heterogeneous Treatment Effects in Two Randomized Controlled Trials. Am J Respir Crit Care Med. 2023 Apr 1;207(7):945-949. doi: 10.1164/rccm.202210-1988LE. No abstract available. PMID 36656551
- [Derived] Kraft R, Herndon DN, Finnerty CC, Shahrokhi S, Jeschke MG. Occurrence of multiorgan dysfunction in pediatric burn patients: incidence and clinical outcome. Ann Surg. 2014 Feb;259(2):381-7. doi: 10.1097/SLA.0b013e31828c4d04. PMID 23511841
- [Derived] Jeschke MG, Williams FN, Finnerty CC, Rodriguez NA, Kulp GA, Ferrando A, Norbury WB, Suman OE, Kraft R, Branski LK, Al-mousawi AM, Herndon DN. The effect of ketoconazole on post-burn inflammation, hypermetabolism and clinical outcomes. PLoS One. 2012;7(5):e35465. doi: 10.1371/journal.pone.0035465. Epub 2012 May 11. PMID 22606232
- [Derived] Jeschke MG, Gauglitz GG, Kulp GA, Finnerty CC, Williams FN, Kraft R, Suman OE, Mlcak RP, Herndon DN. Long-term persistance of the pathophysiologic response to severe burn injury. PLoS One. 2011;6(7):e21245. doi: 10.1371/journal.pone.0021245. Epub 2011 Jul 18. PMID 21789167
- [Derived] Jeschke MG, Kraft R, Emdad F, Kulp GA, Williams FN, Herndon DN. Glucose control in severely thermally injured pediatric patients: what glucose range should be the target? Ann Surg. 2010 Sep;252(3):521-7; discussion 527-8. doi: 10.1097/SLA.0b013e3181f2774c. PMID 20739853
- [Derived] Mecott GA, Herndon DN, Kulp GA, Brooks NC, Al-Mousawi AM, Kraft R, Rivero HG, Williams FN, Branski LK, Jeschke MG. The use of exenatide in severely burned pediatric patients. Crit Care. 2010;14(4):R153. doi: 10.1186/cc9222. Epub 2010 Aug 11. PMID 20701787
- [Derived] Jeschke MG, Kulp GA, Kraft R, Finnerty CC, Mlcak R, Lee JO, Herndon DN. Intensive insulin therapy in severely burned pediatric patients: a prospective randomized trial. Am J Respir Crit Care Med. 2010 Aug 1;182(3):351-9. doi: 10.1164/rccm.201002-0190OC. Epub 2010 Apr 15. PMID 20395554
- [Derived] Gauglitz GG, Herndon DN, Kulp GA, Meyer WJ 3rd, Jeschke MG. Abnormal insulin sensitivity persists up to three years in pediatric patients post-burn. J Clin Endocrinol Metab. 2009 May;94(5):1656-64. doi: 10.1210/jc.2008-1947. Epub 2009 Feb 24. PMID 19240154
- [Derived] Jeschke MG, Chinkes DL, Finnerty CC, Kulp G, Suman OE, Norbury WB, Branski LK, Gauglitz GG, Mlcak RP, Herndon DN. Pathophysiologic response to severe burn injury. Ann Surg. 2008 Sep;248(3):387-401. doi: 10.1097/SLA.0b013e3181856241. PMID 18791359

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients admitted to burn unit with >40% burn or greater
Pre-assignment Details: At the request of the study site, this study has been closed. Access to study-related data is unavailable, and the PI is no longer at the institution. Hence, we are unable to submit the results data. Although peer-reviewed articles have been located that reference NCT00673309, it is not clear and verifiable (without access to the actual study-related data) what the results for the study outcomes are.
Groups:
- Growth Hormone Administration: Growth Hormone administered daily until 95% wound healing. Stable Isotope Infusion Study with collection of blood and tissue
  Stable Isotope Infusion study: Stable isotope infusion study to be done following each surgery. Tagged isotopes to assess uptake into blood and tissues. Includes collection of blood and tissues (muscle)
  Growth Hormone: Recombinant Human Growth hormone to be administered daily until 95% wound healing.
- Insulin High Dose Administration: Insulin IV administered continuously to 95% healing. Stable Isotope Infusion Study with collection of blood and tissue
  Stable Isotope Infusion study: Stable isotope infusion study to be done following each surgery. Tagged isotopes to assess uptake into blood and tissues. Includes collection of blood and tissues (muscle)
  Insulin: Insulin IV administered continuously throughout hospitalization until wounds are 95% healed.
- Oxandrolone Administration: Oxandrolone administered daily until 95% wound healing Stable Isotope Infusion Study with collection of blood and tissue
  Stable Isotope Infusion study: Stable isotope infusion study to be done following each surgery. Tagged isotopes to assess uptake into blood and tissues. Includes collection of blood and tissues (muscle)
  oxandrolone: Oxandrolone given daily throughout hospitalization until 95% wound healing.
- Propranolol Administration: Propranolol administered daily until 95% wound healing Stable Isotope Infusion Study with collection of blood and tissue
  Stable Isotope Infusion study: Stable isotope infusion study to be done following each surgery. Tagged isotopes to assess uptake into blood and tissues. Includes collection of blood and tissues (muscle)
  Propranolol: Propranolol to be given daily throughout hospitalization until 95% wound healing.
- Itraconazole Administration: Itraconazole administered throughout hospitalization until 95% wound healing Stable Isotope Infusion Study with collection of blood and tissue
  Stable Isotope Infusion study: Stable isotope infusion study to be done following each surgery. Tagged isotopes to assess uptake into blood and tissues. Includes collection of blood and tissues (muscle)
  Itraconazole administered throughout hospitalization until 95% wound healing.
- IGF-1/IGFBP-3 Comparator: IGF-1/IGFBP-3 administered daily to 95% wound healing. Stable Isotope Infusion Study with collection of blood and tissue
  Stable Isotope Infusion study: Stable isotope infusion study to be done following each surgery. Tagged isotopes to assess uptake into blood and tissues. Includes collection of blood and tissues (muscle)
  IGF-1/IGFBP-3 administered until 95% wound healing
- Insulin Low Dose Administration: Insulin IV administered continuously through hospitalization to 95% wound healing.
- Growth Hormone and Propranolol Administration: Growth Hormone and Propranolol administration throughout hospitalization to 95% wound healing.
  Includes stable isotope infusion studies.
- Oxandrolone and Propranolol: Oxandrolone and Propranolol administration throughout hospitalization to 95% wound healing.
  Includes stable isotope infusion studies
- Control or Placebo: Control or Placebo administered through hospitalization to 95% wound healing. Includes stable isotope infusion studies.
Period: Overall Study
Arm/Group | Growth Hormone Administration | Insulin High Dose Administration | Oxandrolone Administration | Propranolol Administration | Itraconazole Administration | IGF-1/IGFBP-3 Comparator | Insulin Low Dose Administration | Growth Hormone and Propranolol Administration | Oxandrolone and Propranolol | Control or Placebo
Started | 64 | 14 | 14 | 25 | 18 | 35 | 14 | 13 | 17 | 30
Completed | 64 | 14 | 14 | 25 | 18 | 35 | 14 | 13 | 17 | 30
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: At the request of the study site, this study has been closed. Access to study-related data is unavailable, and the PI is no longer at the institution. Hence, we are unable to submit the results data. Although peer-reviewed articles have been located that reference NCT00673309, it is not clear and verifiable (without access to the actual study-related data) what the results for the study outcomes are.
Groups:
- Total: Total of all reporting groups
Arm/Group | Growth Hormone Administration | Insulin High Dose Administration | Oxandrolone Administration | Propranolol Administration | Itraconazole Administration | IGF-1/IGFBP-3 Comparator | Insulin Low Dose Administration | Growth Hormone and Propranolol Administration | Oxandrolone and Propranolol | Control or Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous
Sex: Female, Male
Protein Net Balance

OUTCOME MEASURES:

1. Primary Outcome: Decrease Hypermetabolism as Measured by Stable Isotope Infusion Study
Description: At the request of the study site, this study has been closed. Access to study-related data is unavailable, and the PI is no longer at the institution. Hence, we are unable to submit the results data. Although peer-reviewed articles have been located that reference NCT00673309, it is not clear and verifiable (without access to the actual study-related data) what the results for the study outcomes are.
Time Frame: Admission to burn unit to 95% wound healing
Population: as for baseline characteristics
Arm/Group | Growth Hormone | Insulin High Dose | Oxandrolone | Propranolol | IGF-1/IGFBP-3 | Insulin Low Dose | Itraconazole | Growth Hormone and Propranolol | Oxandrolone and Propranolol | Control/Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Improved Rate of Wound Healing
Description: as for outcome 1
Time Frame: Admission to burn unit to 95% wound healing
Population: as for baseline characteristics
Arm/Group | Growth Hormone | Insulin High Dose | Oxandrolone | Propranolol | IGF-1/IGFBP-3 | Insulin Low Dose | Itraconazole | Growth Hormone and Propranolol | Oxandrolone and Propranolol | Control/Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Incidence of Morbidity and Mortality
Description: as for outcome 1
Time Frame: Admission to burn unit to discharge
Population: as for baseline characteristics
Arm/Group | Growth Hormone | Insulin High Dose | Oxandrolone | Propranolol | IGF-1/IGFBP-3 | Insulin Low Dose | Itraconazole | Growth Hormone and Propranolol | Oxandrolone and Propranolol | Control/Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Incidence of Sepsis
Description: as for outcome 1
Time Frame: Admission to burn unit to 95% wound healing
Population: as for baseline characteristics
Arm/Group | Growth Hormone | Insulin High Dose | Oxandrolone | Propranolol | IGF-1/IGFBP-3 | Insulin Low Dose | Itraconazole | Growth Hormone and Propranolol | Oxandrolone and Propranolol | Control/Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: At the request of the study site, this study has been closed. Access to study-related data is unavailable, and the PI is no longer at the institution. Hence, we are unable to submit the results data. Although peer-reviewed articles have been located that reference NCT00673309, it is not clear and verifiable (without access to the actual study-related data) what the results for the study outcomes are.
Description: At the request of the study site, this study has been closed. Access to study-related data is unavailable, and the PI is no longer at the institution. Hence, we are unable to submit the results data. Although peer-reviewed articles have been located that reference NCT00673309, it is not clear and verifiable (without access to the actual study-related data) what the results for the study outcomes are.
Groups:
- EG000: unknown - Shriner's Burn Hospital revoked access to study-related data.. We are unable to submit the additional information or results-data.
Arm/Group | EG000
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
At the request of the study site, this study has been closed. Access to study-related data is unavailable, and the PI is no longer at the institution. Hence, we are unable to submit the results data. Although peer-reviewed articles have been located that reference NCT00673309, it is not clear and verifiable (without access to the actual study-related data) what the results for the study outcomes are.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No